CLINICAL TRIAL: NCT04374773
Title: Effect of Estradiol and Cortisol on Marinol Metabolism
Brief Title: Effects of Pregnancy-associated Hormones on THC Metabolism in Women
Acronym: PrECEPT
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Nina Isoherranen, Professor, School of Pharmacy, University of Washington
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: STUDY00008064; 2P01DA032507-06A1 (NIH)
Record Dates: First submitted 2020-04-30; First posted 2020-05-05 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Pregnancy Related; Cannabis Use
Keywords: Pregnancy, cannabis, THC, estradiol, cortisol, women
MeSH Terms: conditions — Marijuana Abuse | interventions — Dronabinol

STUDY DESIGN:
Intervention Model Description: Standard drug-drug interaction study consisting of two arms with randomized, open-label, two period crossover design
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Estradiol (Experimental): 1 week treatment with 0.3 mg/24 hr transdermal estradiol
  Interventions: Drug: Dronabinol
- Cortisol (Experimental): 1 week treatment with 30 mg hydrocortisone daily, administered in 2 divided doses
  Interventions: Drug: Dronabinol

INTERVENTIONS:
Drug: Dronabinol — 2.5 mg PO administered once prior to and once after 1 week of hormone therapy
  Other Names: THC, tetrahydrocannabinol

SUMMARY:
Cannabis use is prevalent among pregnant women, but the effects of use on both the developing fetus and pregnant woman are unknown. Importantly, drug exposure could be influenced by the impact of pregnancy-associated hormones on the metabolism of tetrahydrocannabinol (THC), the main psychoactive component of cannabis. The goal of this study is to determine whether cortisol and estradiol - hormones that rise dramatically during pregnancy - increase the clearance of dronabinol (THC) in reproductive age women to simulate the pregnant state. The collected data will then be used to predict the time course and magnitude of changes in THC metabolism in pregnant women, particularly with gradually increasing estradiol and cortisol concentrations that evolve over the course of pregnancy. The overall objective of this study is to better understand the effects of THC use during pregnancy on the health of the pregnant woman and developing fetus.

DETAILED DESCRIPTION:
Tetrahydrocannabinol (THC) is approved as a medicinal treatment under the trade name dronabinol but is also a drug of abuse when consumed as part of cannabis products. With the legalization of recreational cannabis use and increased use among pregnant women, there is new urgency to understand the dose-exposure relationship for THC, the mechanisms by which THC is eliminated from the body, and the impact of the hormonal milieu of pregnancy on these mechanisms. As approximately 4% of all pregnant women in the United States use cannabis, there is a critical need for studies evaluating how cannabis metabolism may change during pregnancy leading to altered exposures, pharmacology, and toxicology. Recent studies suggest that cannabis exposure during pregnancy may adversely affect the developing fetus, and administration of cannabis [or dronabinol (THC)] to pregnant women is therefore not ethical. Analysis of THC exposures and effects during pregnancy is significantly hindered by the lack of accurate, quantitative biomarkers of THC exposure and the unreliable self-report of cannabis use. To address these gaps, the current study is designed to 1) characterize the dose-exposure relationship of THC and its major metabolites 11-OH-THC and 11-nor-carboxy-THC in reproductive age women following consumption of dronabinol orally and 2) to determine how THC metabolism is altered by the pregnancy-associated hormones estradiol and cortisol. Existing data show that THC and its major metabolites are cleared by metabolizing enzymes whose activity increases during pregnancy and further has been shown to be induced specifically by estradiol and cortisol, hormones that are markedly increased during pregnancy. Based on these data, we hypothesize that increasing estradiol and cortisol concentrations during pregnancy will increase the clearance of THC and its metabolites, leading to an altered metabolism in pregnant women when compared to non-pregnant individuals. Our clinical study seeks to determine the magnitude of changes in THC pharmacokinetics in healthy female volunteers following exposures to increased estradiol and cortisol. We predict that increased estradiol and cortisol concentrations will result in induction of THC-metabolizing enzymes in the liver and intestine, resulting in increased clearance of THC and its metabolites. The clinical study will provide the foundation for modeling and simulation of THC disposition during human pregnancy. These studies will also provide seminal data to allow modeling of the THC metabolome in human plasma and urine as a function of THC dose and time after consumption, making a significant impact on development of reliable biomarkers of THC exposures in humans.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, premenopausal women ages 21-45 years old
* Body mass index (BMI) <30 kg/m2
* Regular menstrual periods (monthly, cycle 28-35 days in length)
* Willingness to use nonhormonal methods of contraception during the study period

Exclusion Criteria:

* History of diabetes or significant cardiac, kidney (eGFR<60 mL/min/1.73m2), gastrointestinal or liver disease
* History of blood clots or stroke
* Allergy to dronabinol, synthetic steroids, or any other chemically related drug or steroid
* Current or recent ingestion (<3 weeks) of any medication or herbal supplement known to be an inducer or inhibitor of CYP2C9, CYP3A4 or UGT. These include some anticoagulants, anti-psychotics, antibiotics, antifungal agents, antidepressants, anti-retroviral agents and herbal supplements (or other over-the-counter medications and supplements). Subjects who are taking any of these prescription drugs will not be asked to discontinue treatment but will be ineligible for study participation. Subjects taking excluded over-the-counter medications and/or supplements will be given the option of discontinuing these for 1 month prior to study participation.
* Current pregnancy or lactation
* History of use of illicit drugs or smoking within the last year
* Any recreational or medicinal use of cannabis or other forms of THC within 3 months
* Current use of amphetamines, anticholinergic drugs or antidepressants
* History of seizure disorder or psychiatric illness (mania or schizophrenia; major depression within the past year or >2 episodes lifetime)
* Current use of live or live attenuated vaccines
* Personal or family (1st degree relative) history of breast or ovarian cancer
* Systemic disease (cancer, auto-immune disease, chronic infection, etc)
* Current or recent (within 6 months) use of hormonal contraceptives
* History of severe hypertriglyceridemia (>300 mg/dL or history of acute pancreatitis)
* Uncontrolled hypertension (BP>140/90)
* Allergy to sesame oil
* Anemia (Hct <34 g/dL)
* Extensive skin disease (eczema, psoriasis, etc) that would preclude use of transdermal estradiol

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2020-10-19 (Actual); Primary Completion 2025-08-14 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Dronabinol exposure | 24 hours
  Area under plasma concentration-time curve (AUC) for THC

SECONDARY OUTCOMES:
THC primary metabolite exposure | 24 hours
  Area under plasma concentration-time curve (AUC) for 11-OH-THC
THC secondary metabolite exposure | 24 hours
  Area under plasma concentration-time curve (AUC) for 11-nor-COOH-THC
Pharmacologic effects of THC | 12 hours
  Visual analog scale ratings of subjective 'high'

CONTACTS AND LOCATIONS:
Overall Officials: Nina Isoherranen, PhD, Principal Investigator — University of Washington
Locations (1):
- Nina Isoherranen, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No